CLINICAL TRIAL: NCT00056004
Title: Phase II Trial Of Zileuton In Persons With Bronchial Dysplasia
Brief Title: Zileuton in Preventing Lung Cancer in Patients With Bronchial Dysplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000271915; P30CA022453 (NIH); WSU-D-2405; WSU-093201MP4F
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Head and Neck Cancer; Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer; stage I non-small cell lung cancer; stage I squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the nasopharynx; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Squamous Cell Carcinoma of Head and Neck | interventions — zileuton

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: zileuton

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of zileuton may be an effective way to prevent lung cancer in patients who have bronchial dysplasia.

PURPOSE: Randomized phase II trial to study the effectiveness of zileuton in preventing lung cancer in patients who have bronchial dysplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of zileuton, in terms of number of sites and grade of dysplastic lesions in the bronchial epithelium, in patients with documented bronchial dysplasia.
* Correlate the regression of bronchial dysplasia (number and grade) and improvement in sputum cytology with the modulation of molecular biomarkers in patients treated with this drug.
* Determine the overall toxicity of this drug in these patients.
* Determine the 6-month natural history of bronchial dysplasia in patients who are randomized to receive treatment with a placebo.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to smoking status (current vs recently quit smoker), and prior cancer (none vs lung or head and neck). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral zileuton 4 times daily for 6 months in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral placebo 4 times daily for 6 months in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL: Approximately 134 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At high risk for dysplasia, defined by 1 of the following criteria:

  * Current or former smokers who have smoked at least 30 pack-years

    * Former smokers must be enrolled within 20 years of complete smoking cessation
  * Patients with curatively treated stage I non-small cell lung cancer*
  * Patients with curatively treated stage I or II squamous cell carcinoma of the head and neck (limited to oral cavity, pharynx, or larynx)* NOTE: *At least 12 months post-curative therapy
* Histologic confirmation of mild to severe bronchial dysplasia on bronchoscopic biopsy required

  * Moderate or severe atypia on sputum cytology required before bronchoscopy (not required for patients with prior lung or head and neck cancer)
* No evidence of malignancy by chest x-ray

PATIENT CHARACTERISTICS:

Age

* 18 and over (for patients with prior lung or head and neck malignancy)
* 35 and over (for all other patients)

Performance status

* SWOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10.0 g/dL
* No bleeding disorder

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* Liver enzymes no greater than ULN
* PT/PTT no greater than ULN
* No active or chronic liver disease (even if transaminases have normalized)

Renal

* Creatinine no greater than ULN

Cardiovascular

* No unstable angina
* No uncontrolled heart failure

Pulmonary

* No significant asthma or chronic obstructive pulmonary disease requiring chronic or periodic (at least once per year) steroids for flares
* No acute or chronic respiratory failure

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing and able to undergo serial bronchoscopic examinations
* No ongoing alcohol use (i.e., at least 1 glass of wine, beer, or a mixed drink per day on a regular basis)
* No other medical condition that would preclude safety during study participation
* No other active or invasive malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix
* No hypersensitivity to study drug or any of its inactive ingredients

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* More than 3 months since prior corticosteroids*
* No concurrent corticosteroids*
* No concurrent anticancer hormonal agents NOTE: *Systemic or inhaled, including chronic administration

Radiotherapy

* No concurrent radiotherapy

Surgery

* Not specified

Other

* More than 3 months since prior lipoxygenase inhibitors*
* More than 3 months since prior investigational agents
* More than 3 months since prior nutritional supplements (except 1 daily multivitamin)
* No concurrent nutritional supplements (except 1 daily multivitamin)
* No other concurrent lipoxygenase inhibitors*
* No other concurrent investigational agents
* No concurrent warfarin, beta-blockers, or theophylline
* No other concurrent antineoplastic agents
* No concurrent or chronic daily use of non-steroidal anti-inflammatory agents (NSAIDS) (except cardioprotective doses of aspirin less than 100 mg/day)

  * Periodic use of NSAIDS allowed
* Concurrent participation in a smoking cessation program (including use of bupropion or nicotine gum or patch) allowed NOTE: *Systemic or inhaled, including chronic administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2003-06; Primary Completion 2006-09 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Bronchial dysplasia number and grade at 6 months

SECONDARY OUTCOMES:
Biomarkers (Ki-67, Cyclin D1, bcl-2, bax, caspase-3) by immunohistochemistry at 6 and 12 months
Biomarkers (5-HETE, LTB-4) by blood and BAL levels at 6 and 12 months
Adverse events as measured by number and severity monthly

CONTACTS AND LOCATIONS:
Overall Officials: Omer Kucuk, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States